CLINICAL TRIAL: NCT03648593
Title: The Effects of Counselling Delivered Through Native Mobile Application on Work Ability and Work Recovery Among Micro-entrepreneurs
Brief Title: Promo@Work Entrepreneurs
Acronym: Promo@Work
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: University of Oulu (Other); Tampere University (Other); University Hospital of Cologne (Other); Academy of Finland (Other)
Responsible Party: Principal Investigator, Jaana Laitinen, Chief Specialist, Principal Investigator, PhD,, Finnish Institute of Occupational Health
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 3522101; 303430 (Other Grant/Funding Number: Strategic Research Council at the Academy of Finland)
Record Dates: First submitted 2018-05-24; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Work Ability; Work-Related Condition; Health Behavior; Intervention
Keywords: microenterpreneur; work ability; work recovery; native mobile app; health behaviour; work; stress; work performance
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: randomized intervention trial with waiting list control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- behavioral (Experimental): work recovery intervention
  Interventions: Behavioral: work recovery intervention
- waiting list control (Experimental): work recovery intervention after 6 months
  Interventions: Behavioral: waiting list control

INTERVENTIONS:
Behavioral: work recovery intervention — Recover! app: one hour weekly for two months
  Arms: behavioral
Behavioral: waiting list control — no treatment during 6 months,then Recover! app
  Arms: waiting list control

SUMMARY:
A randomized intervention study to promote work recovery and work ability among micro-entrepreneurs. The main aim is to investigate if the use of Recovery! -application results in better work recovery and work ability than no treatment for micro-entrepreneurs.

The plan of action of the study merges: 1) the contents that are based on the needs of the target population and evidence from research on work related and health behaviour enhancing work recovery, 2) theoretical framework for the counselling, 3) counselling methods including behaviour change techniques, and 4) tailoring the content and counselling according to trans theoretical change model and physical work demands. The intervention is delivered through native mobile application designed by using the abovementioned methodology.

Data are collected by repeated internet-based questionnaires (at baseline, 2 and 6 months from the beginning of the intervention) and from the use of mobile application. Furthermore, randomly selected persons in two groups (20-30 persons in each) are interviewed. Process evaluation is conducted to detect the mechanisms of change and to study why the program succeeded or failed.

ELIGIBILITY:
Inclusion Criteria:

* Finnish-speaking micro-entrepreneurs (those with enterprise of 1-9 employees),
* company is located in Finland.
* work full-time as entrepreneurs,
* understand Finnish,
* use an Android phone.

Exclusion Criteria:

* not full-time entrepreneurs
* on sick leave
* absent from work

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1256 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-08-30 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline in need for recovery scale at 6 months | change from baseline in need for recovery scale at 6 months
  need for recovery scale measures early symptoms of fatigue
change from baseline in perceived work ability at 6 months. One item of work ability index | change from baseline in perceived work ability at 6 months
  to rate their work ability on a scale of 0 to 10, ten being their lifetime best work ability

SECONDARY OUTCOMES:
change from baseline in 3-item version of the Utrecht Work Engagement Scale at 6 months | change from baseline in 3-item version of the Utrecht Work Engagement Scale at 6 months
  "At my work, I feel bursting with energy" (vigor); (2) "I am enthusiastic about my job"(dedication);(3)"I am immersed in my work" (absorption)
Change from baseline in Recovery Experiences Questionnaire at 6 months | change from baseline in Recovery Experiences at 6 months
  The Recovery Experience Questionnaire - a Measure for assessing recuperation and unwinding from work
World health organization Health and work performance questionnaire | change from baseline in work performance at 6 months
  World health organization Health and work performance questionnaire
sleep deprivation questions | change from baseline in sleep deprivation at 6 months
  Sleep deprivation is calculated by subtracting hours slept from hours of sleep needed
Frequency of insomnia symptoms | change from baseline in insomnia symptoms at 6 months
  Symptoms of insomnia are difficulties falling asleep, waking up at nights, waking up too early in the morning unable to fall asleep again and feeling of sleep which does not refresh. How often have you had this kind of symptoms during last 3 months?" Answers were given using Likert-scale: 1) Never or less than once a month, 2) less than once a week, 3) 1-2 days a week, 4) 3-5 days a week or 5) daily or almost daily.
nutritional behaviour | change from baseline in nutritional behaviour at 6 months
  number of meals and snacks per day
Alcohol Use Disorders Identification Test Consumption (Audit-C) | change from baseline in Audit-C at 6 months
  the Finnish version of the questionnaire Alcohol Use Disorders Identification Test Consumption 3 questions
physical activity questionnaire | change from baseline in physical activity at 6 months
  frequency in light and brisk physical activities (daily, four to six times a week, two to three times a week, once a week, two to three times a month, and once a month or less often). The duration of one bout of activity was considered separately for light and brisk activities (over 90 minutes, 60 to 90 minutes, 40 to59 minutes, 20 to 39 minutes, less than 20 minutes, and not at all)

OTHER OUTCOMES:
dose of intervention | from baseline until 2 months
  dose of Recover application (using time in hours and minutes during two months)

CONTACTS AND LOCATIONS:
Overall Officials: Jaana Laitinen, PhD, Docent, Principal Investigator — Chief Specialist
Locations (1):
- Finnish Institute of Occupational Health, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kekkonen M, Korkiakangas E, Laitinen J, Oinas-Kukkonen H. Factors Reducing the Use of a Persuasive mHealth App and How to Mitigate Them: Thematic Analysis. JMIR Hum Factors. 2023 Jun 26;10:e40579. doi: 10.2196/40579. PMID 37358883